CLINICAL TRIAL: NCT01798550
Title: Evaluation of Enoxaparin Dosing in Hospitalized Morbidly Obese Patients at an Academic Medical Center
Brief Title: Enoxaparin Dosing in Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Christine Kempton, MD, MSc, Associate Professor, Department of Pediatrics and Department of Hematology and Medical Oncology, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00063210
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-10

CONDITIONS: Obesity
Keywords: Enoxaparin dosing; Obesity
MeSH Terms: conditions — Obesity | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reduced Dose (0.8 mg/kg) (Experimental): Enoxaparin 0.8 mg/kg (using total body weight) twice daily
  Interventions: Drug: Enoxaparin
- Standard Dose (1 mg/kg) (Active Comparator): Enoxaparin 1 mg/kg (using total body weight) twice daily
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Twice daily dosing
  Other Names: Lovenox

SUMMARY:
The purpose of this study is to determine an effective enoxaparin dosing strategy in medically ill, morbidly obese patients. This study will include adult patients greater than 18 yrs of age being admitted to Grady Hospital in Atlanta, GA. Potentially vulnerable patients such as prisoners, children, and pregnant women will not be enrolled in the study. Study participants will be contacted in person by the study personnel once inclusion criteria are met. Written informed consent will be obtained in person while hospitalized. Once the patient is consented they will be given enoxaparin and blood samples will be drawn. The data collected will be from the electronic medical record which is accessed only with a username and password so it is not publicly available. The data will be identifiable upon collection and will be kept on a password protected file on a computer in a locked office. The data will be de-identified after data analysis and only the study personnel will have access to the code that links identifiers to subjects. A HIPAA waiver will be requested to access existing data in order to identify patients for enrollment. All data will be collected in an office in the hospital. The study participants' burden will be minimal and dependent only on time of consent process since morbidly obese patients would be receiving this blood sample collection regardless of their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Planned treating with twice daily enoxaparin
* BMI >= 40 kg/m2

Exclusion Criteria:

* < 18 years of age
* CrCl < 30 ml/min
* Pregnancy
* Prisoner
* Active bleeding
* Already received 3 consecutive doses of enoxaparin
* Use of therapeutic enoxaparin for more than 5 consecutive days within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-03; Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine L Kempton, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reduced Dose (0.8 mg/kg) | Standard Dose (1 mg/kg)
Started | 30 | 32
Completed | 28 | 26
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reduced Dose (0.8 mg/kg) | Standard Dose (1 mg/kg) | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Median (Full Range); unit: years] | 55 [45 to 62] | 56 [46 to 63] | 56 [45 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 30
  Male | 18 | 14 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 27 | 54
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With an Initial Therapeutic Anti-Xa Level at Steady State in Each Group
Time Frame: 3-5 hours after at least 3rd dose
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Dose (0.8 mg/kg) | Standard Dose (1 mg/kg)
Number analyzed (Participants) | 28 | 26
Participants | 25 | 20

2. Secondary Outcome: Time to Therapeutic Anti-Xa Level for Both Groups
Description: Time to therapeutic Anti-Xa = time in hours from enoxaparin dose #1 to the first therapeutic Anti-Xa. The Anti-Xa was assessed 3-5 hours after at least three consecutive enoxaparin doses. If a dose adjustment was needed, the anti-Xa level was drawn four hours after the adjusted dose of enoxaparin was administered. Dose adjustments were made until a therapeutic level within goal range was obtained.
Time Frame: Assessed once after 3 consecutive enoxaparin doses (approx. 36 hours) and then daily if dose adjustments were indicated up to 30 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Reduced Dose (0.8 mg/kg) | Standard Dose (1 mg/kg)
Number analyzed (Participants) | 28 | 26
hours | 28.6 [26.7 to 41.0] | 31.9 [27.7 to 39.2]

3. Other Pre Specified Outcome: Median Steady State Anti-Xa Levels
Description: The goal anti-Xa peak level range was defined as 0.5 - 1.1 International units/mL. The Anti-Xa was assessed 3-5 hours after at least three consecutive enoxaparin doses. If a dose adjustment was needed, the anti-Xa level was drawn four hours after the adjusted dose of enoxaparin was administered. Dose adjustments were made until a therapeutic level within goal range was obtained.
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: IU/mL
Arm/Group | Reduced Dose (0.8 mg/kg) | Standard Dose (1 mg/kg)
Number analyzed (Participants) | 28 | 26
IU/mL | 0.8 [0.66 to 0.90] | 0.86 [0.69 to 1.01]

4. Other Pre Specified Outcome: Number of Patients Requiring Dose Adjustments to Achieve Therapeutic Anti-Xa Level
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Dose (0.8 mg/kg) | Standard Dose (1 mg/kg)
Number analyzed (Participants) | 28 | 26
Participants | 3 | 6

5. Other Pre Specified Outcome: Proportion of Patients With Major and Minor Bleeding Events Prior to Achieving a Therapeutic Level
Time Frame: Hemoglobin and platelets were assessed at baseline and daily as indicated while on study up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Dose (0.8 mg/kg) | Standard Dose (1 mg/kg)
Number analyzed (Participants) | 28 | 26
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years, duration of the study
Arm/Group | Reduced Dose (0.8 mg/kg) | Standard Dose (1 mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 0/30 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT01798550/Prot_SAP_000.pdf